CLINICAL TRIAL: NCT00804557
Title: Efficacy And Safety Of The Uro-Ease® Urinary Catheter During Clean Intermittent Catheterization
Status: Terminated | Type: Observational
Why Stopped: pending design changes to the device
Sponsor: Lahey Clinic (Other)
Collaborators: Spirus Medical, Inc. (Industry)
Responsible Party: John T. Stoffel, M.D., Lahey Clinic, Inc.
Other Study IDs: 2008-065
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Urinary Retention; Urinary Catheterization
Keywords: Male Urinary Disorders; Urinary catheterization; Urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Uro-Ease Spirus Catheter: 10 patients randomized to the Uro-Ease Catheter group for 1 week. In clinic, patients will be instructed in the use of the Uro-Ease Catheter. A QOL form will be filled out measuring comfort and ease of use and subsequently after each catheterization. Patients will also record time per catheterization and bladder drainage. Patients will return to Clinic in 1 week to check progress and will then change to a standard, non-helical urinary catheter. Patients will be followed up to 1 month.
- Standard Urinary Catheter: 10 patients randomized to a Standard Urinary Catheter group for 1 week. In clinic, patients will be instructed in the use of the catheter. A QOL form will be filled out measuring comfort and ease of use and subsequently after each catheterization. Patients will also record time per catheterization and bladder drainage. Patients will return to Clinic in 1 week to check progress and will then change to the UroEase Spirus Catheter. All patients will be followed up to 1 month.

SUMMARY:
To evaluate the ease of use and comfort of a new urinary catheter, the Uro-Ease, as used in the Clean Intermittent Catheterization (CIC)process.

DETAILED DESCRIPTION:
Urinary retention can occur among men with Benign Prostatic Hypertrophy(BPH) or Neurologic co-morbidities.

Many of these men are treated with Clean Intermittent Catheterization(CIC. For some, this can be a time consuming and often painful process due to difficulty with catheter insertion and manipulation, which may result in urethral injury or non-compliance.

The blunt nose of a standard catheter can meet significant resistance at the external sphincter or within the prostate urethra. Spirus Medical has developed a urinary catheter, Uro-Ease, with a rounded helical thread formed on the surface of its distal end for use in CIC.

This study is to determine whether the design of the Uro-Ease catheter allows for easier Clean Intermittent self-Catheterization(CIC) while maintaining safe bladder drainage.

This is a prospective randomized study with two phases.

Phase 1: Observational, 5 patients. In this phase, five patients meeting the inclusion criteria will be consented from the Urology Clinic. Participating Urology nurses who have been previously trained in the utilization of the Spirus Catheter, will perform the initial CIC on the patient with a 12 Fr Spirus Catheter(choice of 2 different flexibilities). The study nurse will document time per catheterization and effective drainage of bladder. Before leaving the clinic, patient's will be instructed in the use of the Spirus Catheter and demonstrate efficacy with using the Spirus Catheter. Patients will then fill out VAS Forms for ease and comfort of catheter insertion and after each subsequent catheterization. Patients will also record, for 3 consecutive days, time it takes for catheterization and time to drain the bladder . Patients will return to clinic in 1 week to return VAS forms and documentation. A follow-up phone call will be made to the patient in month to check on patient's status.

All patients will be instructed to call clinic, nurse or on-call-urologist for any report of urethral trauma, which will be evaluated with flexible cystoscopy. These reports will be reviewed and documented.

Phase 2: Randomized crossover trial, 20 patients. After successful completion of Phase 1, patients will be randomized into 2 groups-10 patients will first be randomized into the Spirus Catheter Group and 10 patients into the Standard 12 FR Bard Catheter Group.(Coude' or straight catheters may be utilized for standard group) As in Phase 1, all patients will receive CIC instruction for self-catheterization, specific to the selected catheter and can demonstrate efficacy with CIC using selected catheter, before they leave the clinic. Patients will then fill out VAS forms for catheter insertion ease and comfort and after each subsequent catheterization. Patient will also record time per catheterization and bladder drainage for 3 consecutive days. Patients will return to the clinic in 1 week for a progress report, return VAS forms and reports. At this time the patient will be switch over to the alternate catheter group for 1 week.

All patients will be instructed to call clinic, nurse or on-call-urologist for any report of urethral trauma, defined as blood on catheter or per meatus. Any occurence of urethral trauma will be evaluated with flexible cystoscopy. These reports will be reviewed and documented.

All patients will be followed up to one month to check on the patient's status.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Urinary retention defined as >150cc retained in bladder on post void residual

Exclusion Criteria:

* Female patients
* Known urethral stricture
* Active symptomatic Urinary Tract Infection
* History of pelvic fracture or urethral disruption
* History of previous urethroplasty(urethral reconstructive surgery)
* Known Latex allergy
* Unable to physically perform CIC
* Unable to provide follow up
* Unable to give consent
* Currently taking chronic narcotic pain medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from Lahey Clinic Urology Service and colleague referrals
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine whether the design of the Uro-Ease Catheter device allows for easier, more comfortable clean intermittent self-catheterization (CIC) while maintaining safe bladder drainage. Using Visual Analog Scales and Timed procedure logs | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John T. Stoffel, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Kashefi C, Messer K, Barden R, Sexton C, Parsons JK. Incidence and prevention of iatrogenic urethral injuries. J Urol. 2008 Jun;179(6):2254-7; discussion 2257-8. doi: 10.1016/j.juro.2008.01.108. Epub 2008 Apr 18. PMID 18423712
- [Background] Logan K, Shaw C, Webber I, Samuel S, Broome L. Patients' experiences of learning clean intermittent self-catheterization: a qualitative study. J Adv Nurs. 2008 Apr;62(1):32-40. doi: 10.1111/j.1365-2648.2007.04536.x. PMID 18352962
- [Background] Jahn P, Preuss M, Kernig A, Seifert-Huhmer A, Langer G. Types of indwelling urinary catheters for long-term bladder drainage in adults. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004997. doi: 10.1002/14651858.CD004997.pub2. PMID 17636782
- [Background] Webb RJ, Lawson AL, Neal DE. Clean intermittent self-catheterisation in 172 adults. Br J Urol. 1990 Jan;65(1):20-3. doi: 10.1111/j.1464-410x.1990.tb14653.x. PMID 2310927
- [Background] Woodward S, Rew M. Patients' quality of life and clean intermittent self-catheterization. Br J Nurs. 2003 Oct 9-22;12(18):1066-74. doi: 10.12968/bjon.2003.12.18.11782. PMID 14581839
- [Background] Shaw C, Logan K, Webber I, Broome L, Samuel S. Effect of clean intermittent self-catheterization on quality of life: a qualitative study. J Adv Nurs. 2008 Mar;61(6):641-50. doi: 10.1111/j.1365-2648.2007.04556.x. PMID 18302605
- [Background] Liedberg H. Catheter induced urethral inflammatory reaction and urinary tract infection. An experimental and clinical study. Scand J Urol Nephrol Suppl. 1989;124:1-43. PMID 2633310
- [Background] Ferrie BG, Groome J, Sethia B, Kirk D. Comparison of silicone and latex catheters in the development of urethral stricture after cardiac surgery. Br J Urol. 1986 Oct;58(5):549-50. doi: 10.1111/j.1464-410x.1986.tb05465.x. PMID 3490896
- [Background] Bull E, Chilton CP, Gould CA, Sutton TM. Single-blind, randomised, parallel group study of the Bard Biocath catheter and a silicone elastomer coated catheter. Br J Urol. 1991 Oct;68(4):394-9. doi: 10.1111/j.1464-410x.1991.tb15359.x. PMID 1933160
- [Background] Erickson BA, Navai N, Patil M, Chang A, Gonzalez CM. A prospective, randomized trial evaluating the use of hydrogel coated latex versus all silicone urethral catheters after urethral reconstructive surgery. J Urol. 2008 Jan;179(1):203-6. doi: 10.1016/j.juro.2007.08.174. Epub 2007 Nov 14. PMID 18001794